CLINICAL TRIAL: NCT00363298
Title: Double-blind Trial of Acute and Intermediate-term Dextro-amphetamine Versus Caffeine Augmentation in Treatment Resistant Obsessive Compulsive Disorder (OCD)
Brief Title: Dextro-Amphetamine Versus Caffeine in Treatment-resistant OCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Obsessive Compulsive Foundation (Other)
Responsible Party: Principal Investigator, Lorrin M Koran, Professor of Psychiatry, Emeritus, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 97134
Record Dates: First submitted 2006-08-09; First posted 2006-08-15 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-02

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: D-amphetamine, dextro-amphetamine, stimulant drug
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Dextroamphetamine; Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- d-amphetamine (Experimental): dextro-amphetamine capsules, 15 mg per capsule, in Bottles A and B, dose: one from Bottle A each morning and 1 from Bottle B each morning
  Interventions: Drug: dextro-amphetamine
- Sham comparison (Sham Comparator): caffeine in capsules identical to those containing d-amphetamine, with 200 mg of caffeine in Bottle A capsules, and 100 mg of caffeine in Bottle B capsules, dose was 1 capsule from Bottle A and 1 capsule from Bottle B each morning
  Interventions: Drug: Sham Comparison

INTERVENTIONS:
Drug: dextro-amphetamine — dextro-amphetamine dosage form: 15 mg capsules, in Bottles A and B. Dosage: One capsule from Bottle A and one capsule from bottle B each morning. Frequency: once daily. Duration: 5 weeks.
  Other Names: Dexedrine
  Arms: d-amphetamine
Drug: Sham Comparison — caffeine dosage form: capsules identical to those in dextro-amphetamine arm, but containing 200 mg caffeine in Bottle A and 100 mg caffeine in Bottle B. Frequency: once daily. Duration: 5 weeks
  Other Names: Caffeine, 300 mg/day
  Arms: Sham comparison

SUMMARY:
The study hypothesis is that dextro-amphetamine (d-amphetamine) will be safe and effective when used to augment treatment for Obsessive-Compulsive Disorder (OCD), and that tolerance (loss of therapeutic effect) to the medication will not develop over a period of several weeks.

DETAILED DESCRIPTION:
The study will investigate whether dextro-amphetamine (d-amphetamine) is safe and effective compared to caffeine as an active placebo when used to augment treatment for Obsessive-Compulsive Disorder (OCD), and whether tolerance (loss of therapeutic effect) to the medication will develop over a period of several weeks

D-amphetamine is approved by the U.S. Food and Drug Administration to treat Attention Deficit Hyperactivity Disorder (ADHD) in children and adolescents. Because of the effects that d-amphetamine has on the brain, Dr. Koran believes it may be helpful in treating OCD. A positive finding in this study may stimulate research aimed at improving OCD treatment and understanding of the neurochemistry involved.

This research study will enroll 24 people who are taking medication for their OCD but are not receiving sufficient benefit. The research will be performed only at Stanford University.

ELIGIBILITY:
Inclusion Criteria:

* outpatient age 18 through 55 inclusive
* meets DSM-IV criteria for obsessive-compulsive disorder (OCD) with Yale-Brown Obsessive-Compulsive Scale (YBOCS) score greater than or equal to 20
* provides written informed consent
* has taken for at least 12 weeks at least the dose shown of a selective serotonin reuptake inhibitor (SSRI) [citalopram, escitalopram, or fluoxetine 20 mg/d; paroxetine 40 mg/d; sertraline 50 mg/d]; or venlafaxine 225 mg/d; or duloxetine 60 mg/d.
* if taking buspar, gabapentin, an atypical antipsychotic, or a benzodiazepine, dose has been stable for 4 weeks
* has negative urine drug and pregnancy tests
* is practicing reliable birth control method
* has blood pressure readings at screening visit that are less than 140 mm Hg systolic and 90 mm Hg diastolic,
* weight is greater than 100 lbs at screen

Exclusion criteria:

* requires psychotropic medications other than an Serotonin Reuptake Inhibitor (SRI), a benzodiazepine, buspirone, an atypical antipsychotic, and/or gabapentin
* is taking clomipramine
* is taking fluvoxamine
* is taking medication that inhibits hepatic enzyme CYP1A2
* is taking a monoamine oxidase inhibitor
* has co-morbid tics or Tourette's disorder
* has hoarding as the primary or only OCD symptom
* has a history of panic disorder
* has a history of glaucoma
* has a history of seizures
* has a history of schizophrenia or psychotic disorder, or schizotypal personality disorder
* has depression with current suicide risk
* has mental retardation, pervasive developmental disorder, or cognitive disorder
* has a factitious disorder
* has current or past cyclothymic disorder or bipolar disorder
* has a dissociative disorder
* has personality disorder sufficient to interfere with study participation
* has organic mental disorder or dementia
* has current or past substance abuse / dependence (excluding nicotine)
* has current or past anorexia or bulimia
* has serious or unstable medical disorder, including hypertension or cardiac disease
* has history of myocardial infarction or cardiac arrhythmia
* has history of or has current diagnosis of hypertension
* is pregnant or breast-feeding
* is receiving psychotherapy for OCD
* is intending to receive psychotherapy for OCD during the study
* has had a previous trial of d-amphetamine of at least 30 days duration
* is unable to speak, read, or understand English
* is not likely to follow study procedures
* is not suitable for study in the investigator's opinion

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2006-08; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorrin M Koran, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Koran LM, Aboujaoude E, Gamel NN. Double-blind study of dextroamphetamine versus caffeine augmentation for treatment-resistant obsessive-compulsive disorder. J Clin Psychiatry. 2009 Nov;70(11):1530-5. doi: 10.4088/JCP.08m04605. Epub 2009 Jun 30. PMID 19573497

RESULTS

PARTICIPANT FLOW:
Groups:
- D-amphetamine: Dextro-amphetamine dosage form: 15 mg capsules, in Bottles A and B. Dosage: One capsule from Bottle A and one capsule from bottle B each morning. Frequency: once daily. Duration: 5 weeks.
  Caffeine dosage form: 200 mg capsules in Bottle A, 100 mg capsules in Bottle B. Dosage: One capsule from Bottle A and one capsule from bottle B each morning. Frequency: once daily. Duration: 5 weeks.
- Caffeine Pills: Caffeine in capsules identical to those containing d-amphetamine, with 200 mg of caffeine in Bottle A capsules, and 100 mg of caffeine in Bottle B capsules. Dose was 1 capsule from Bottle A and 1 capsule from Bottle B each morning. Frequency: once daily. Duration: 5 weeks
Period: First Study Week
Arm/Group | D-amphetamine | Caffeine Pills
Started | 12 | 12
Completed | 6 (At end of week 1, 6/12 subjects met Y-BOCS response criterion and began 4-week continuation phase) | 7 (At end of week 1, 7/12 subjects met Y-BOCS response criterion and began 4-week continuation phase)
Not Completed | 6 | 5
Not completed — Lack of Efficacy | 6 | 5
Period: 4-week Study Continuation Phase
Arm/Group | D-amphetamine | Caffeine Pills
Started | 6 | 7
Completed | 5 | 7
Not Completed | 1 | 0
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Population: 24 Subjects meeting the listed entry criteria.
Groups:
- D-amphetamine: Dextro-amphetamine: dextro-amphetamine dosage form: 15 mg capsules, in Bottles A and B. Dosage: One capsule from Bottle A and one capsule from bottle B each morning. Frequency: once daily. Duration: 5 weeks.
  Caffeine dosage form: 200 mg capsules in Bottle A, 100 mg capsules in Bottle B. Dosage: One capsule from Bottle A and one capsule from bottle B each morning. Frequency: once daily. Duration: 5 weeks.
- Total: Total of all reporting groups
Arm/Group | D-amphetamine | Caffeine Pills | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean Age, and standard deviation, in years
  years
    Baseline Age | 42.3 (12.8) | 37.8 (13.7) | 40.05 (13.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24
Prior Selective Serotonin Reuptake or Serotonin Norepinephrine Reuptake Inhibitor trials [Mean (Standard Deviation); unit: trials] | 3.0 (NA) — Standard deviation was not calculated and the raw data are no longer available | 3.7 (NA) — Standard deviation was not calculated and the raw data are no longer available. | 3.4 (NA) — Standard deviation was not calculated and the raw data are no longer available.
Atypical antipsychotic drug augmentation trials [Mean (Standard Deviation); unit: trials] | 2.4 (NA) — Standard deviation was not calculated and the raw data is no longer available. | 2.5 (NA) — Standard deviation was not calculated and the raw data is no longer available. | 2.5 (NA) — Standard deviation was not calculated and the raw data is no longer available.

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Clinical Global Impressions Scale - Improvement (CGI-I) Score of 1 or 2
Description: Clinical Global Impressions Scale Improvement Score = 1 (very much improved), or 2 (much improved). Additional possible scale scores are 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (much worse) and 7 (very much worse).
Time Frame: At end of week 5, except 1 d-amphetamine subject rated at end of week 2
Population: Subjects who met the study continuation phase entry criterion of >20% decrease in Y-BOCS score after 1 week of double-blind study medication, and entered this 4-week double-blind continuation phase
Measure: Number; unit: participants
Arm/Group | D-amphetamine | Caffeine Pills
Number analyzed (Participants) | 6 | 7
participants | 6 | 7

2. Primary Outcome: Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) Score
Description: Yale-Brown Obsessive-Compulsive Scale score by blinded investigator in direct interview. The scale score is the sum of ten items (5 for obsessions and 5 for compulsions: time occupied, degree of interference with functioning, degree of distress, effort to resist the symptom, success in resisting), each rated from 0 to 4, with higher scores indicating more severe OCD. Maximum score is 40. Scores of 14 and below are often described as "subclinical," though patients with these scores may still exhibit troubling symptoms and mild to moderate distress. A total score of 8 or less is often termed "remission." A decrease in total score from baseline to endpoint of either 25% or 35% is often used as a "responder" criterion in clinical trials.
Time Frame: At end of week 5, except 1 d-amphetamine subject rated at end of week 2
Population: Subjects who entered the 4-week double-blind study continuation phase, including a last observation carried forward for the one d-amphetamine subject who dropped out of this phase at the end of study week 2 (end of the first week of the continuation phase) for lack of efficacy.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-amphetamine | Caffeine Pills
Number analyzed (Participants) | 6 | 7
units on a scale | 13.3 (6.9) | 13.0 (8.4)

ADVERSE EVENTS:
Time Frame: 1 week for 11 subjects who did not meet entry criteria for the 4-week extension phase, 2 weeks for the single subject who discontinued in week 2 for lack of efficacy and 5 weeks for the 12 subjects who completed the extension phase.
Groups:
- D-amphetamine: Dextro-amphetamine dosage form: 15 mg capsules, in Bottles A and B. Dosage: One capsule from Bottle A and one capsule from bottle B each morning. Frequency: once daily. Duration: 5 weeks.
Arm/Group | D-amphetamine | Caffeine Pills
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 5/12 | 4/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | D-amphetamine (N=12) | Caffeine Pills (N=12)
insomnia (Psychiatric disorders) | 2 | 2
dry mouth (Gastrointestinal disorders) | 2 | 0
decreased appetite (Gastrointestinal disorders) | 1 | 0
nausea (Gastrointestinal disorders) | 0 | 1
intermittent jitteriness (Nervous system disorders) | 0 | 1
Decrease in drug dose (Blood and lymphatic system disorders) | 3 | 1 — non-sustained increase in pulse or systolic blood pressure
Irritability (Psychiatric disorders) | 0 | 1 — irritability

LIMITATIONS AND CAVEATS:
Modest sample size of 24 subjects, 12 in each drug group. Observation period was only 5 weeks long.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No